CLINICAL TRIAL: NCT03045484
Title: Comparison of Controlled-release Oxycodone to Control Chemoradiotherapy-induced Moderate or Severe Oral Mucositis Pain in Nasopharyngeal Carcinoma Patients
Brief Title: Comparison of Oxycodone to Control Moderate or Severe Oral Mucositis Pain Induced by Chemoradiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ling Guo, Principal Investigator;Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2015-058-01
Record Dates: First submitted 2016-10-31; First posted 2017-02-07 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: nasopharyngeal carcinoma; Oral Mucositis Pain; Oxycodone
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Chemoradiotherapy; Radiotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The moderate group (Experimental): Patient who was suffering from moderate pain in the mouth, pharynx, or larynx during the treatment of chemoradiotherapy consented to take controlled-release oxycodone, oxycodone was begun at the level of mild pain. We called this the moderate group. Controlled-release oxycodone was used to relieve oral mucositis pain induced by chemoradiotherapy in this group.
  Interventions: Drug: Controlled-release oxycodone; Other: Chemoradiotherapy
- The severe group (Experimental): Patients who did not ask for controlled-release oxycodone until the pain reached a moderate level during the treatment of chemoradiotherapywere called the severe group. Controlled-release oxycodone was also used to relieve oral mucositis pain induced by chemoradiotherapy in this group..
  Interventions: Drug: Controlled-release oxycodone; Other: Chemoradiotherapy

INTERVENTIONS:
Drug: Controlled-release oxycodone — CRO is effective for 12 h. Patient takes it only twice a day. The minimum oral unit of CRO is a 10 mg tablet, so the minimum daily dose was 10 mg.
  Other Names: CRO
Other: Chemoradiotherapy — Radiotherapy were administered intensity modulated radiation therapy wiht a dose of 1.8-2.2Gy per fraction, 30-32 fraction for various tumor locations. Chemotherapy drugs platinum was used once a weak with 100mg/㎡.
  Other Names: Radiotherapy and Chemotherapy

SUMMARY:
Background:Although concurrent chemoradiotherapy is effective for improving disease-free survival and overall survival in patients with locally advanced nasopharyngeal carcinoma. However,the oral mucositis pain evoked by the chemoradiotherapy itself reduces food intake and frequently halts the treatment. Thus, pain control is an important problem in chemoradiotherapy for nasopharyngeal carcinoma.We performed to examine whether early induction of low-dose, opioid from moderate pain reduced total dose of Oxycodone during chemoradiotherapy, while improves the quality of life and reduce weight loss.

Objective:Present clinical trial to investigate the early introduction of opioids suppressed the transient increase in the numeric rating scales(NRS) score for pain and compared with conventional treatment.

Methodology:The subjects will recruit 70 patients who were hospitalized for nasopharyngeal carcinoma. 70 patients were divided into two groups, depending on whether the pain was moderate or severe when an opioid was introduced.Differences between groups were compared using T test protected least significant difference for one-factor analysis of variance. All statistical analyses were performed using SPSS(Statistic Package for Social Science) software.P-values < 0.05 were considered statistically significant.

DETAILED DESCRIPTION:
Controlled-release oxycodone (CRO) was used in this study. The patients kept a daily record of the intensity of pain. CRO is effective for 12 h, so that the patient takes it only twice a day.The minimum oral unit of CRO is a 10 mg tablet, so the minimum daily dose was 20 mg. Thus, we began at a dose of 20 mg by default. When the pain worsened, the dose was quickly titrated.When a patient who was suffering from moderate pain in the mouth, pharynx, or larynx consented to take oxycodone, oxycodone was begun at the level of moderate pain. We called this the mild group. In contrast, those patients who did not ask for oxycodone until the pain reached a severe level were called the severe group. Because all patients agreed to use an opioid at some point, the patients were classified into two groups, moderate and severe, according to when the opioid was introduced.

Total dose of oxycodone was defined as the total dose of oxycodone taking during the treatment of chemoradiotherapy. Pain Remission Rate was defined as pain remission after 24h from the start of opioid administration.Evaluating quality of life were conducted once every two weeks.We also evaluated the weight loss as parameters for food intake once a week,until the radiotherapy.All statistical analyses were performed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18 to 65 years.

  * Patients of both genders must be willing to practice birth control from the time of enrollment on this study.
  * Participants with treatment- Chemoradiotherapy advanced Nasopharyngeal carcinoma.
  * Participants with the ability to assess the pain level.
  * Never use a opioid before treatment.
  * Hematology:

WBC≥4.0×109/L, ANC≥1.5×109/L, PLT≥100×109/L,Hb≥90g/L.

Exclusion Criteria:

* •Patients do not conform to the inclusion criteria.

  * Refuse to use of opioid drugs.
  * Nasopharyngeal patients with mental illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Total Dose of Oxycodone | Through chemoradiotherapy completion, 3 weeks

SECONDARY OUTCOMES:
Pain Remission Rate | 24 hours
Quality-of-Life Index | Through chemoradiotherapy completion, an average of 2 weaks

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guo SP, Wu SG, Zhou J, Feng HX, Li FY, Wu YJ, Sun JY, He ZY. Transdermal fentanyl for pain due to chemoradiotherapy-induced oral mucositis in nasopharyngeal cancer patients: evaluating efficacy, safety, and improvement in quality of life. Drug Des Devel Ther. 2014 May 12;8:497-503. doi: 10.2147/DDDT.S60187. eCollection 2014. PMID 24872680
- [Background] Takase H, Sakata T, Yamano T, Sueta T, Nomoto S, Nakagawa T. Advantage of early induction of opioid to control pain induced by irradiation in head and neck cancer patients. Auris Nasus Larynx. 2011 Aug;38(4):495-500. doi: 10.1016/j.anl.2010.12.012. Epub 2011 Jan 31. PMID 21277720
- [Background] Lauretti GR, Oliveira GM, Pereira NL. Comparison of sustained-release morphine with sustained-release oxycodone in advanced cancer patients. Br J Cancer. 2003 Dec 1;89(11):2027-30. doi: 10.1038/sj.bjc.6601365. PMID 14647133
- [Background] Epstein JB, Epstein JD, Epstein MS, Oien H, Truelove EL. Management of pain in cancer patients with oral mucositis: follow-up of multiple doses of doxepin oral rinse. J Pain Symptom Manage. 2007 Feb;33(2):111-4. doi: 10.1016/j.jpainsymman.2006.11.002. No abstract available. PMID 17280915